CLINICAL TRIAL: NCT06038500
Title: Effect of an Intervention of Dance, Resistance Exercises and Nutritional Recommendations on Muscle Mass and Strength in Women With Risk of Sarcopenia
Brief Title: Multicomponent Intervention in Women at Risk of Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: University of Guadalajara (Other); Universidad de Colima (Other)
Responsible Party: Principal Investigator, Maria Claudia Espinel Bermudez, Principal Investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R-2019-1310-040
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Sarcopenia; Grip Strength; Gait Speed; Body Composition
Keywords: Sarcopenia; Multicomponent; Aging; Preventive
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: quasi-experimental Pre-test/Post-test design - pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicomponent Intervention in only one group of women at Risk of Sarcopenia (Experimental): Quasi-experimental Pre-test/Post-test design - pilot
  Interventions: Other: Multicomponent intervention of resistance exercises, dancing sessions and nutritional education

INTERVENTIONS:
Other: Multicomponent intervention of resistance exercises, dancing sessions and nutritional education — The intervention consisted of two sets of ten repetitions of resistance exercises, the second month four sets of eight repetitions, and the third month four sets of fifteen repetitions. It was estimated that each session (dance + resistance exercise) generated a caloric expenditure of 270.85 calories corresponding to 4.5 and 3.5 METs per activity. The resistance exercises and the dance sessions began and with a warm-up and stretching session 10 min, followed by the resistance exercises 30 min and dancing practice 30 min. The session ended with a cooling down session 10 min. The nutritional education offered included weekly topics lasting 20 min, on basic concepts of nutrition and recommended diet for the maintenance of skeletal muscle mass. Reinforcement of the topics was carried out through triptychs that were provided throughout the 12 sessions.

SUMMARY:
The goal of this quasi-experimental pilot study is to evaluate the effect of a multi-component intervention in women between 55 and 75 years old at risk of sarcopenia. The main question it aims to answer are: What is the effect of a multi-component intervention in women at risk of sarcopenia? Participants will twelve women between 55 and 75 years old with risk of sarcopenia, who agreed through written informed consent for participate 12 weeks with 24 sessions included dancing, resistance exercises, and nutritional education. The outcomes were muscle mass, grip strength, gait speed and body composition. The effects were measured before and after the intervention, under a self-controlled design.

DETAILED DESCRIPTION:
Physical exercise, especially resistance exercise, is one of the best non-pharmacological treatment alternatives due to its multiple health benefits and could be a promoter for the prevention of sarcopenia by delaying muscle atrophy produced by the natural aging process. However, scientific literature shows that this activity when combined with other strategies has a better effect on sarcopenia indicators than alone. Dance is a social activity that is part of the culture and life history of human beings, however, current research has focused on studying the cognitive and visuospatial effects of this activity. It could be an activity with beneficial effects on the physical abilities of the individual since dancing improves flexibility, resistance and balance. However, the study of these two strategies, along with nutritional education has been little studied.

Therefore, a pilot test was proposed with the aim of knowing the possible effect of a multicomponent intervention on muscle, strength, performance, and body composition on women at risk of sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Positive requested through written informed consent
* Current public health insurance
* Preserved physical and mental capacities (verified through data from the medical record)
* Having a lower grip strength, less or equal to 20.99 kg
* Appendicular skeletal muscle index (ASMI) maintained, greater or equal to 5.5 kg/m^2
* Walking speed greater or equal to 0.8 m/s

Exclusion Criteria:

* Bioelectric activity add (osteosynthesis metal systems or devices, pacemakers, defibrillators)
* Alterations of body composition (history of cancer, uncontrolled chronic degenerative diseases, risk of malnutrition, respiratory insufficiency, asthma or chronic obstructive pulmonary disease, hospitalization in the year prior to the study; limitations in carrying out the basic activities of daily living; medical contraindication for physical activity, and or belonging to another physical activity group).

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Grip strength | Baseline measurement and final measurement as the end of the 12 weeks of intervention
  Evaluated with the JAMAR Plus+ Patterson Medical® digital dynamometer, using the technique proposed by the American Society of Hand Therapists. It was based on the average among all the attempts done on each hand. The results were obtained in kilograms (kg).
Skeletal muscle mass index (SMI) | Baseline measurement and final measurement as the end of the 12 weeks of intervention
  Based on the formula validated by Yamada et al (10.3390/ijerph14070809) for multi-frequency devices using the measurements taken with a TANITA MC 780 (ALM = (0.6947 × (Ht^2/Z50)) + (-55.24 × (Z250/Z5)) + (-10,940 × (1/Z50)) + 51.33)
Gait speed | Baseline measurement and final measurement as the end of the 12 weeks of intervention
  Evaluated with a stopwatch to estimate the time after acceleration and before deceleration for a total distance of 4 meters. The unit of measurement was meters between seconds (m/s).

SECONDARY OUTCOMES:
Anthropometric measurements | Baseline measurement and final measurement as the end of the 12 weeks of intervention
  Height, mid-arm, waist, hip, and calf measurements stipulated by the ISAK protocol, all measurements were quantified in centimeters (cm).

OTHER OUTCOMES:
Polypharmacy report (yes/no) | Baseline measurement
  Obtained direct information of women about current pharmacological regimens for diseases. Polypharmacy was defined as the use of five or more medications according to what was established by Integrated care for older people (ICOPE) of the WHO.
Comorbidity | Baseline measurement
  Obtained direct information of women about diseases assessed using the Charlson index.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Claudia Espinel-Bermudez, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Rios-Escalante V, Perez-Barba JC, Espinel-Bermudez MC, Zavalza-Gomez AB, Arias-Merino ED, Zavala-Cerna MG, Sanchez-Garcia S, Trujillo X, Nava-Zavala AH. Effects of a Multicomponent Preventive Intervention in Women at Risk of Sarcopenia: A Pilot Study. Healthcare (Basel). 2024 Jun 13;12(12):1191. doi: 10.3390/healthcare12121191. PMID 38921304